CLINICAL TRIAL: NCT04776109
Title: Analgesic Efficacy of Erector Spinae Infusion Versus Thoracic Epidural Infusion of Bupivacaine for Postoperative Pain in Patients Undergoing Upper Abdominal Cancer Surgeries
Brief Title: Analgesic Efficacy of Erector Spinae Infusion Versus Thoracic Epidural for Patients With Upper Abdominal Cancer Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Hussein Mahmoud, assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 521
Record Dates: First submitted 2021-02-18; First posted 2021-03-01 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Pain Relief in Upper Abdominal Cancer Surgeries

STUDY DESIGN:
Intervention Model Description: First group (Group of continous thoracic epidural bupivacaine infusion [CEI]) Second group (Group of continous bilateral erector spinae bupivacaine infusions[CESI])
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- (Group of continous thoracic epidural bupivacaine infusion [CEI]) (Active Comparator): Group I : An epidural catheter will be inserted via a paramedian approach as close as possible to the surgical procedure via the inter-vertebral space (from T8 to T10) so that the affected dermatomes of the surgical wound would receive the benefits of bupivacaine (sunny-bupivacaine) infusion. Proper placement of the catheter will be verified through an aspiration test and a test dose (2 ml) of lidocaine 2% with adrenaline. At the end of surgery, a 0.2 ml/kg bolus of bupivacaine 0.25% will be administered through the catheter and then an infusion of bupivacaine 0.125% at a rate of 0.1 ml/kg/h will be administered immediately postoperative and continued for 48 hours.
  Interventions: Procedure: erector spinae block
- (Group of continous bilateral erector spinae bupivacaine infusions[CESI]) (Active Comparator): Group II : Bilateral erector spinae catheters will be placed at T8 level. Surface anatomy or ultrasound (counting up from the 12th rib) will be used to identify the level of T8 after skin sterilization with the patient on the lateral position. Then a high frequency linear-array ultrasound transducer (Sono Site MW, Bothell, WA, USA) covered in a sterile sleeve will be placed in a longitudinal parasagittal orientation 3 cm lateral to the midline to identify the back muscles: the trapezius above, the rhomboid major in the middle, and the erector-spinae muscle on the bottom, and the transverse Processes with shimmering pleura in between. Next, 2-3 ml of 2% lidocaine will be infiltrated. A catheter will be inserted and secured. The procedure will be repeated on the contralateral side. 20 ml of bupivacaine 0.25% solution will be injected immediately into each catheter then infusion of bupivacaine 0.125% 0.1 ml/kg/h will be continued for 48 hours.
  Interventions: Procedure: erector spinae block

INTERVENTIONS:
Procedure: erector spinae block — Bilateral erector spinae catheters will be placed at T8 level. an ultrasound transducer will be placed in a longitudinal parasagittal orientation 3 cm lateral to the midline to identify the back muscles and the transverse Processes. Next, 2-3 ml of 2% lidocaine will be infiltrated .
  A 16-G, 8-cm Tuohy needle will be then introduced medially in the plane of the ultrasound beam and directed towards the transverse process. Once the needle is underneath the anterior fascia of the erector spinae muscle, 10 ml of saline 0.9% will be injected lifting the muscle of the transverse process. A catheter will be inserted into the newly formed space underneath the ES muscle and secured. The procedure will be repeated on the contralateral side. bupivacaine (20 ml of bupivacaine 0.25%) solution will be injected immediately into each catheter then infusion of bupivacaine 0.125% 0.1 ml/kg/h will be continued for 48 hours.
  Other Names: thoracic epidural block

SUMMARY:
Epidural analgesia is considered by many to be the reference standard which has been shown to reduce the intraoperative surgical stress response.

However, besides its excellent analgesic effect, there are some disadvantages associated with epidural analgesia. This includes the risk of epidural hematoma/abscess ,failure rates hypotension, urinary retention. Also the need for preoperative placement in awake patients, who seem to dislike and sometimes even refuse. It is contra-indicated in the presence of coagulopathy or local sepsis.

ESPB is a faster procedure that carries a lower risk of hypotension, can be used in patients with coagulopathy, easy to perform, and requires less training.

So this study is to compare the postoperative analgesic effect of continous bupivacaine infusion via thoracic epidural versus erector spinae catheters following upper abdominal cancer surgery.

DETAILED DESCRIPTION:
Surgical trauma activates numerous receptors leading to severe postoperative pain. Therefore, effective pain management is a priority of care and a patient right.

Postoperative pain may cause tachycardia, hypertension, increased cardiac work, nausea, vomiting, ileus. Also if it is inadequately managed may lead to detrimental Cardiovascular effects, pulmonary dysfunction, immune system, neuro-endocrine and metabolic effects, gastrointestinal, urinary dysfunction, coagulation system , cognitive dysfunction and also have psychological, economic and social adverse effects Good postoperative analgesia can prevent morbidity associated with abdominal surgeries by allowing pain-free, early ambulation and decreasing the risks of long hospital stay, thromboembolism, and other poor outcomes.

Adequate pain treatment is an important component of modern perioperative care and essential for a fast recovery. Choosing the optimal analgesic modality remains a topic of debate especially in major abdominal surgeries.

Epidural analgesia is considered by many to be the reference standard. It is used routinely in many thoracic surgery centers. Epidural blockade has been shown to reduce the intraoperative surgical stress response and has possible advantages for cardiovascular, respiratory, coagulation, gastrointestinal, metabolic and immune function However, besides its excellent analgesic effect, there are some disadvantages associated with epidural analgesia. This includes the risk of epidural hematoma/abscess (incidence 1:1,000-6,000 in surgical patients), failure rates of up to 30%, hypotension, urinary retention , in rare cases; paraplegia. Also the need for preoperative placement in awake patients, who seem to dislike and sometimes even refuse . It is contra-indicated in the presence of coagulopathy or local sepsis.

In the last decade, there has been a significant shift away from thoracic epidural analgesia (TEA) that has been long considered as the gold standard.

Various techniques have been tried to replicate the analgesic efficacy of TEA. They include transversus abdominis plane analgesia (TAP), rectus sheath analgesia (RS), wound infusion analgesia (WI) and transmuscular quadratus lumborum (TQL) analgesia.

However each of these techniques has specific limitations that prevent them from being the analgesic technique of choice for all open abdominal surgeries.

Epidural analgesia is commonly used in patients following abdominal surgeries except in cases with elevated intracranial tension, coagulopathy, patient refusal, and local sepsis.

Truncal blocks such as transversus abdominis plane (TAP) blocks have seen limited success due to shorter duration and suboptimal analgesia.

The ultrasound (US)-guided erector spinae plane block (ESPB) was initially described by Forero et al.It as a relatively new technique, originally described to manage thoracic pain when performed at the T5 vertebra level, but it has also been successfully used for abdominal analgesia when performed at T7 level.

ESPB gained wide attention as it is a faster procedure that carries a lower risk of hypotension, can be used in patients with coagulopathy, easy to perform, and requires less training.

ESPB provides extensive, potent unilateral analgesia, performed by local anesthetic injection in the plane between the erector spinae muscle and the TP. The local anesthetic diffuses into the paravertebral space through spaces between adjacent vertebrae and blocks both the dorsal and ventral rami of the thoracic spinal nerves.

Bilateral ESPB performed at low thoracic levels provides satisfactory analgesia for abdominal surgeries in case reports and series describing abdominal exploration, cesarean section, ventral hernia repair, and abdominoplasty. [21-23] As LA widely spreads cranially and caudally when ESPB is performed, we think that ESPB can effectively be used as an analgesic method for abdominal surgeries.

Aims of the study The objective of this study is to compare the postoperative analgesic effect of continous bupivacaine infusion via thoracic epidural versus erector spinae catheters following upper abdominal cancer surgery

Patients and Methods After obtaining institutional ethical committee approval and written informed consent from each patient, patients undergoing major upper abdominal cancer surgery who will be applicable to our study inclusion criteria ( at South Egypt Cancer Institute from December 2020 to December 2022) will be enrolled in this study.

patients will be randomized by the use of computer generated table of random numbers in a 1:1 ratio and conducted using a numbered, opaque and sealed envelope into two groups, First group (Group of continous thoracic epidural bupivacaine infusion [CEI]) Second group (Group of continous bilateral erector spinae bupivacaine infusions[CESI]) Group I : An epidural catheter will be inserted via a paramedian approach as close as possible to the surgical procedure via the inter-vertebral space (from T8 to T10) so that the affected dermatomes of the surgical wound would receive the benefits of bupivacaine (sunny-bupivacaine) infusion. Proper placement of the catheter will be verified through an aspiration test and a test dose (2 ml) of lidocaine 2% with adrenaline. At the end of surgery, a 0.2 ml/kg bolus of bupivacaine 0.25% will be administered through the catheter and then an infusion of bupivacaine 0.25% at a rate of 0.1 ml/kg/h will be administered immediately postoperative and continued for 48 hours.

Group II : Bilateral erector spinae catheters will be placed at T8 level. Surface anatomy or ultrasound (counting up from the 12th rib) will be used to identify the level of T8 after skin sterilization with the patient on the lateral position. Then a high frequency linear-array ultrasound transducer (Sono Site MW, Bothell, WA, USA) covered in a sterile sleeve will be placed in a longitudinal parasagittal orientation 3 cm lateral to the midline to identify the back muscles: the trapezius above, the rhomboid major in the middle, and the erector-spinae muscle on the bottom, and the transverse Processes with shimmering pleura in between. Next, 2-3 ml of 2% lidocaine will be infiltrated .

A 16-G, 8-cm Tuohy needle (Portex; Smiths Medical International Ltd, Kent, UK) will be then introduced medially in the plane of the ultrasound beam and directed towards the transverse process. Once the needle is underneath the anterior fascia of the erector spinae muscle, 10 ml of saline 0.9% will be injected. The injectate will be observed spreading underneath the ES muscle lifting the muscle of the transverse process. A catheter (Portex; Smiths Medical International Ltd) will be inserted into the newly formed space underneath the ES muscle and secured. The procedure will be repeated on the contralateral side. bupivacaine (20 ml of bupivacaine 0.25%) solution will be injected into each catheter over five minutes and then an infusion of bupivacaine 0.25% at a rate of 0.1 ml/kg/h will be administered immediately postoperative and continued for 48 hours on both sides.

Postoperatively, all patients will receive IV morphine (3 mg) when needed with VAS score < 3 for a period of 48 hours.

Procedures will be done under complete antiseptic technique. General anesthesia In the preoperative room, standard monitoring probes will be attached, IV 18 G cannula will be inserted and 1 L of normal saline will be infused. In the operative room, after pre-oxygenation for 3 minutes, anesthesia will be induced with intravenous (propofol 1.5 mg/kg) and fentanyl 2 μg/kg. Tracheal intubation will be performed after adequate neuromuscular blockade with rocuronium 0.6 mg/kg. Anesthesia will be maintained by isoflurane 1-1.5 MAC, rocuronium 0.3 mg/kg will given when indicated. Fentanyl 0.5 μg/kg will be given to maintain heart rate (HR) and blood pressure within 20% of the basal value. Patients will be mechanically ventilated to maintain end tidal (ETCO2) between 35-40 mmHg. The inspired oxygen fraction (FIO2) will be 0.5 using oxygen-and-air mixtures. At the end of surgery neuromuscular block will antagonized in all patients with sugammadex 1μg/kg and finally the patients will be extubated in the operative room. Hypotension will determined as a systolic blood pressure < 85 mmHg and will be managed with IV ephedrine 0.1 mg/kg. Bradycardia will be determined as heart rate slower than 50 beats/min and will be given atropine 0.01 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

* Patients subjected to major upper abdominal cancer surgery.
* The enrolled age will be from 18 years to 70 years
* ASA I-II and NYHA I-II.

Exclusion Criteria:

* ASA physical status >II, and NYHA >II
* Patient refusal
* body mass index >40 kg/m2
* preoperative opioid consumption
* a local infection at the incision site
* a history of hematological disorders or coagulation abnormality
* previous abdominal surgeries, severe hepatic or renal impairment
* Anomalies of vertebral column.
* Pregnant women
* Hypersensitivity to any of used drugs
* chronic pain

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
pain intensity measured by 11 points Visual Analogue Scale | immediately postoperative for 48 hours after surgery.
  to assess pain intensity at rest and during pain-provoking movements (deep breathing, coughing, mobilization) measured by 11 points Visual Analogue Scale (VAS) score in which 0 indicates no pain and 10 indicates the severest pain

SECONDARY OUTCOMES:
Hemodynamic variable measured by blood pressure in mmHG | immediately postoperative for 48 hours after surgery.
Hemodynamic variable measured by heart rate in beats per minute | immediately postoperative for 48 hours after surgery.

OTHER OUTCOMES:
total opioid consumption | during first 48 hours postoperatively.
  by measuring total morphine given in mg

CONTACTS AND LOCATIONS:
Locations (1):
- South Egypt Cancer Institute, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided